CLINICAL TRIAL: NCT03692793
Title: Short, Medium and Long-term Effects of Pulmonary Rehabilitation in Dyspnea, Health Status, Anxiety and Depression Symptoms, Functional Status and Postural Control and Its Relationship With Morbimortality in Patients With COPD
Brief Title: Pulmonary Rehabilitation in Functional Outcomes and Its Relationship With Morbidity and Mortality in Patients With COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the Covid-19 pandemic, face-to-face activities have been suspended since March 2020, making the research unfeasible.
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Prof. Dra. Anamaria Fleig Mayer, Principal Investigator, University of the State of Santa Catarina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NuReabPRP
Record Dates: First submitted 2018-09-16; First posted 2018-10-02 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Minimal Clinically Important Difference; Exercise Test; Rehabilitation; Disability Evaluation; Activities of Daily Living; Motivation; Self-efficacy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary rehabilitation (Experimental): The PRP (24-session, three times for week) will be delivered according to ATS/ERS (Spruit et al, 2013),
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — Patients will perform continuous aerobic training (treadmill walking) during 30min (60% of the 6MWT mean speed) and progression according to dyspnea (4-6 of the modified Borg scale). Upper limbs resistance training will be performed using the modified diagonals from the proprioceptive neuromuscular facilitation method (2 sets of 2min). Lower limbs strength training will be performed for quadriceps and triceps sural (2 sets of 10 repetitions), with progression when the patients report that the exercise are ´easy´. All the muscle exercised and the breathing accessory muscles will be stretched for 30s. Eleven educational sessions will be delivered addressing topics related to COPD self-management.

SUMMARY:
Background: The pulmonary rehabilitation effects on various outcomes of COPD are well known. However, they may be lost over time due to poor adherence to therapy with absence of regular exercise maintenance in long term, disease progression, comorbidities, falls incidence and higher exacerbations frequency. Currently, the main focus is to make the patient more active and ensure the benefits maintenance. However, few studies have been concerned with the aim of to investigate the long-term effect of this intervention and the relationship of the change promoted in important outcomes of the disease with its morbidity and mortality.

Design: Non-controlled clinical trial, prospective and longitudinal. Setting: Outpatient pulmonary rehabilitation program in Florianopolis, Brazil

Subjects: Patients with COPD (GOLD II-IV).

Interventions: Pulmonary rehabilitation program (PRP) based on physical training, conducted over 24 sessions supervised, three times a week, including aerobic training in treadmill and resistance training for upper and lower limbs.

Main measures: Before, post-PRP, 6 months post-PRP and 12 months post-PRP will be measured Spirometry or Total Body Plethysmography, Triaxial Accelerometry by Dynaport Activity Monitor, Glittre ADL-Test to evaluated functional capacity and functional performance, Six-Minute Walk Test distance on tracks of 20 and 30 meters, muscle oxygenation variables by NIRS PortaLite®, force platform NeuroCom® SMART Equitest®, Timed Up and Go Test, Berg Balance Scale, Activities-specific Balance Confidence, Falls Efficacy Scale - International - Brasil, London Chest Activity of Daily Living score, Modified Medical Research Council score, Saint George Respiratory Questionnaire score, COPD Assessment Test score and Hospital Anxiety and Depression Scale, Behavioural Regulation in Exercise Questionnaire-2, Basic Psychological Needs in Exercise Scale, General self-efficacy scale, COPD self-efficacy scale, Pulmonary Rehabilitation Adapted Index of Self-Efficacy. The death cases and numbers of exacerbations and hospitalizations will be measured by monthly phone calls after PRP.

DETAILED DESCRIPTION:
Assigned Interventions: Pulmonary rehabilitation program (PRP) will be conducted according to the American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines. Physical training will be conducted over 24 sessions supervised, three times a week. The program will include aerobic training in treadmill (with 30 min load determined by the dyspnea sensation - 4 to 6 on the modified Borg scale) and resistance training for upper limbs with free weights or elastic bands (movements performed based on the proprioceptive neuromuscular facilitation diagonals, performed in two series, lasting two minutes each) and lower limbs (quadriceps and triceps sural) with free weights and/or in the bodybuilding station. All the muscle exercised and the breathing accessory muscles will be stretched for 30s each. Eleven 30-minute educational sessions will be delivered addressing topics related to disease self-management.

The death cases and numbers of exacerbations and hospitalizations will be measured by monthly phone calls after PRP.

Before PRP, post-PRP, 6 months post-PRP and 12 months post-PRP will be evaluated:

Pulmonary function test: Spirometry (EasyOne, NDD) or Total Body Plethysmography (Eric Jaeger, Germany) will be performed in accordance with ATS/ERS standards in order to provide the level of pulmonary obstruction and severity of disease. The predicted values will be calculated with the equations derived from Brazilian population.

Triaxial Accelerometry by Dynaport Activity Monitor: In order to evaluate the physical activity in daily life (PADL), it will be used DynaPort Activity Monitor (McRoberts BV®, Netherlands). Monitoring took place on four consecutive days lasting 12 hours from awakening. Data processing and analysis will be performed with the Dyrector software (McRoberts BV®).

Glittre-ADL Test (TGlittre): The patients will be instructed to complete the circuit described by Skumlien et al. In one day, the patients will perform two Glittre-ADL Tests with the orientation of performing the test in the shortest possible time. On the other day, two tests will also be performed, however, the patients will be instructed to perform the circuit at his usual speed (TGlittre-Perf). The order of execution of TGlittre and TGlittre-Perf will be randomized previously.

Six minute walk test (6MWT): The patients will be instructed to walk in order to perform the largest distance during six minutes. The walking speed will be selected by the patient, according to the guidelines of the ATS. Two 6MWTs will be conducted on tracks of 20 and 30 meters, in different days, with execution order randomized previously.

Peripheral muscle oxygenation: The patients will use a near-infrared spectroscopy device (NIRS PortaLite®, Artinis Medical Systems) on the vastus lateralis muscle of the dominant lower limb during TGlittre, TGlittre-Perf and 6MWT. The positioning will follow the SENIAM Project (Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles) recommendations. The analyzed variables will be oxyhemoglobin, deoxyhemoglobin, total hemoglobin and tissue saturation index.

Postural control: The patients will perform five protocols randomized previously on force platform NeuroCom® SMART Equitest® (Sensory Organization Test, Adaptation Control Test, Motor Control Test, Limits of Stability, Rhythmic Weight Shift e Weight Bearing Squat). Besides, they will perform two Timed Up and Go Test in the shortest possible time and Berg Balance Scale, composed of 14 specific items with different tasks. The Activities-specific Balance Confidence and Falls Efficacy Scale - International - Brasil, both composed for 16 items related to ADL confidence and self-efficacy for falls, respectively, also will be performed. The postural control assessment will be randomized previously.

London Chest Activity of Daily Living scale: Patients will be asked about their perception of limitation in activities of daily living, using the London Chest Activity of Daily Living scale. It consists of 15 items with scores from 0 to 5, with the total score ranging from 0 to 75 points. The higher the score is, the greater the ADL limitation.

Modified Medical Research Council scale: Patients will be asked about their perception of dyspnea, using the modified Medical Research Council scale. The scale range is from 0 to 5, being that higher values correspond to worse dyspnea.

Saint George Respiratory Questionnaire: Patients will be asked about their perception of health-related quality of life, using the Saint George Respiratory Questionnaire. The SGRQ score ranges from 0 to 100% (total and three domains: symptoms, activity and impact), being that higher values correspond to worse quality of life.

COPD Assessment Test: Patients will be asked about the perception of the impact of COPD (cough, sputum, dyspnea, and chest tightness) on health status, using COPD Assessment Test. The total score varies from 0 to 40 and higher scores indicate greater impact of the disease on the health status of these patients.

Hospital Anxiety and Depression Scale: The Hospital Anxiety and Depression Scale will be applied to evaluated symptoms of anxiety and depression. It has two subscales: anxiety and depression. Each subscale generates a final score ranging from 0 to 21 points. Higher scores to more symptoms.

Behavioural Regulation in Exercise Questionnaire-2 (BREQ-2): the questionnaire assesses motivation to exercise. It consists of 19 Likert-based items that measure motivation to exercise. The self-determination index (SDI) will be scored. It ranges between -24 (lowest SDI) to 20 (highest SDI). The higher the SDI score, the greater the motivation to exercise.

Basic Psychological Needs in Exercise Scale: it assesses the patient´s perception regarding the supply of basic psychological needs and with the exercise. It is composed by 12 items that are divided into three domains: autonomy (four items), competence (four items), and relatedness (four items). Each item varies from from 1 ("totally disagree") to 5 ("very strongly agree"). The domains scores varies from 4 to 20. The higher the score, the greater the fulfillment of basic psychological needs.

COPD self-efficacy scale: the scales will be used to assess disease-specific self-efficacy. It assesses an individual's confidence in managing dyspnoea or other breathing-related issues. It is a Likert-based scale, consisting of 34 items divided into the following 5 subscales: negative affect (12 items), intense emotional arousal (8 items), physical exertion (5 items), weather or environment (6 items), behavioural risk factors (3 items). The total score ranges from 34 to 170 points. It can be also presented by a mean of the 34 items (sum of the items divided for 34). The higher the score, the greater the self-efficacy for both scales.

General self-efficacy scale: the scales will be used to assess general self-efficacy. It is a 10-item Likert-based scale, whose score varies from 10 to 40. The higher the score, the greater the self-efficacy.

Pulmonary Rehabilitation Adapted Index of Self-Efficacy: the scale will assess self-efficacy in the context of PR. It is composed by 10 items from the General Self-efficacy Scale and 5 items specific to challenges faced by patients attending a pulmonary rehabilitation program. Each item is scored from 1 to 4, with 4 being the highest level of perceived self-efficacy and 1 being considered the lowest level. The score range comprises a score of 15 to 60, with higher scores indicating high levels of self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD confirmed by spirometry (COPD GOLD stages II, III and IV);
* Clinical stability in the past four weeks.

Exclusion Criteria:

* Hospital admission in the past 12 weeks;
* Any other disease or health condition that could compromise the test´s execution or physical training;
* Participation in pulmonary rehabilitation program completed in the last six months;
* Current smoking or its cessation in less than six months;
* Interruption of pulmonary rehabilitation program for any reason;
* Any change in symptoms during the study protocol assessments.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Physical activity in daily life | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in physical activity in daily life monitoring by accelerometry
Morbidity | Every month after the PRP up to 24 months
  Relationship of changes in outcomes with exacerbation, hospitalization and death
Mortality | Every month after the PRP up to 24 months
  Relationship of changes in outcomes with death

SECONDARY OUTCOMES:
Dyspnea | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  modified Medical Research Council (mMRC) scale. The scale range is from 0 to 5, being that higher values correspond to worse dyspnea
Health status - COPD Assessment Test (CAT) | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  The CAT questionnaire range is from 0 to 40 points (8 items that range from 0 to 5 points each), being that higher values correspond to worse health status
Health status - Saint George Respiratory questionnaire (SGRQ) | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  The SGRQ range is from 0 to 100% (total and three domains: symptoms, activity and impact), being that higher values correspond to worse quality of life
Anxiety and depression symptoms - Hospital Anxiety and Depression Scale (HADS) | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  The HADS range is from 0 to 42 points (two domains: anxiety and depression - 21 points each), being that higher values correspond to more symptoms
Functional status - Glittre-ADL Test (TGlittre) | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in TGlittre
Functional status - Six-Minute Walk Test (6MWT) | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in 6MWT
Functional status - London Chest Activity of Daily Living (LCADL) | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in LCADL. The total score of LCADL (LCADLtotal) range is from 0 to 75 points and the percentage of total score of LCADL (LCADL%total) is calculated by excluding the questions answered zero. As higher the LCADLtotal and LCADL%total scores, worse the functional status
Postural balance - force platform NeuroCom (COP) | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change center of pressure (COP) displacement
Postural balance - force platform NeuroCom (COG) | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in center of gravity (COG) displacement
Postural balance -Timed Up and Go (TUG) Test | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in TUG Test
Postural balance - Berg Balance Scale (BBS) | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in BBS. The scale presents 14 tasks, being that the score range is from 0 to 56 points (from 0 to 4 for each task). As lower the score, worse the postural control
Postural balance - Activities-specific Balance Confidence (ABC) | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in ABC. The scale range is from 0 to 1600% (16 items which range from 0 to 100% each), being that as higher the score, higher the confidence
Postural balance - Falls Efficacy Scale - International - Brasil (FES-I-Brasil) | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in FES-I-Brasil. The scale range is from 0 to 64 (16 items which range from 0 to 4 points each), being that as higher the score, higher the worries about falls
Peripheral muscle oxygenation during exercise and activities of daily living (oxyhemoglobin) | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in oxyhemoglobin of NIRS PortaMon
Peripheral muscle oxygenation during exercise and activities of daily living (deoxyhemoglobin) | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in deoxyhemoglobin of NIRS PortaMon
Peripheral muscle oxygenation during exercise and activities of daily living (total hemoglobin) | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in total hemoglobin of NIRS PortaMon
Peripheral muscle oxygenation during exercise and activities of daily living | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change tissue saturation index of NIRS PortaMon
Motivation - Amotivation | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in amotivation to exercise practice will be assessed by the Behavioural Regulation in Exercise Questionnaire-2 (BREQ-2). Amotivation is scored with the sum of items 5,9,12,19 divided by 4. The score ranges between 0-4 (units on a scale). The higher the score, the greater the amotivation to exercise.
Motivation - External regulation | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in external regulation to exercise practice will be assessed by the Behavioural Regulation in Exercise Questionnaire-2 (BREQ-2). External regulation is scored with the sum of items 1,6,11,16 divided by 4. The score ranges between 0-4 (units on a scale). The higher the score, the greater the external regulation to exercise.
Motivation - Identified regulation | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in identified regulation to exercise practice will be assessed by the Behavioural Regulation in Exercise Questionnaire-2 (BREQ-2). Identified regulation is scored with the sum of items 3,8,14,17 divided by 4. The score ranges between 0-4 (units on a scale). The higher the score, the greater the identified regulation to exercise.
Motivation - Introjected regulation | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in introjected regulation to exercise practice will be assessed by the Behavioural Regulation in Exercise Questionnaire-2 (BREQ-2). Introjected regulation is scored with the sum of items 2,7,13 divided by 3. The score ranges between 0-4 (units on a scale). The higher the score, the greater the external introjected regulation to exercise.
Motivation - Intrinsic regulation | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in intrinsic regulation to exercise practice will be assessed by the Behavioural Regulation in Exercise Questionnaire-2 (BREQ-2). Intrinsic regulation is scored with the sum of items 3,8,14,17 divided by 4. The score ranges between 0-4 (units on a scale). The higher the score, the greater the intrinsic regulation to exercise.
Motivation - Self determination | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in self determination to exercise practice will be assessed by the Behavioural Regulation in Exercise Questionnaire-2 (BREQ-2). Self-determination index (SDI) will be scored based on the equation: [(-3x amotivation)+(-2x external regulation)+(-1x introjected regulation)+(2x identified regulation)+(3x intrinsic regulation). It ranges between -24 (lowest SDI) to 20 (highest SDI). The higher the SDI score, the greater the motivation to exercise.
General Self-efficacy | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in general self-efficacy to exercise assessed by the General self-efficacy scale. The score varies from 10 to 40. The higher the score, the greater the self-efficacy
Disease-specific self-efficacy | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in disease-specific self-efficacy to exercise assessed by the COPD self-efficacy scale. The score ranges from 34 to 170 points. It can be also presented by a mean of the 34 items (sum of the items divided for 34). The higher the score, the greater the self-efficacy for both scales.
Pulmonary Rehabilitation self-efficacy | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in pulmonary-rehabilitation related self-efficacy to exercise assessed by the Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE). The score range comprises a score of 15 to 60, with higher scores indicating high levels of self-efficacy
Basic Psychological Needs | baseline, post-24 sessions of PRP, six months post-PRP, 12 months post-PRP and 24 months post-PRP
  Change in basic psychological needs assessed by the Basic Psychological Needs in Exercise Scale (BPNES). The domains scores (autonomy, competence and relatedness) varies from 4 to 20. The higher the score, the greater the fulfillment of basic psychological needs.

CONTACTS AND LOCATIONS:
Overall Officials: Anamaria F Mayer, PhD, Study Director — University of the State of Santa Catarina
Locations (1):
- Núcleo de Assistência, Ensino e Pesquisa em Reabilitação Pulmonar, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The authors declared that will be shared: individual deidentified participant data; individual data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices); Study Protocol, Statistical Analysis Plan, Informed Consent Form; immediately following publication and ending 5 years following article publication; With Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose to achieve aims in the approved proposal; proposals should be directed to anamaria.mayer@udesc.br to gain access.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: immediately following publication and ending 5 years following article publication
Access Criteria: With Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose to achieve aims in the approved proposal; proposals should be directed to anamaria.mayer@udesc.br to gain access.

REFERENCES:
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Pereira CA, Sato T, Rodrigues SC. New reference values for forced spirometry in white adults in Brazil. J Bras Pneumol. 2007 Jul-Aug;33(4):397-406. doi: 10.1590/s1806-37132007000400008. English, Portuguese. PMID 17982531
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Garrod R, Bestall JC, Paul EA, Wedzicha JA, Jones PW. Development and validation of a standardized measure of activity of daily living in patients with severe COPD: the London Chest Activity of Daily Living scale (LCADL). Respir Med. 2000 Jun;94(6):589-96. doi: 10.1053/rmed.2000.0786. PMID 10921765
- [Background] Carpes MF, Mayer AF, Simon KM, Jardim JR, Garrod R. The Brazilian Portuguese version of the London Chest Activity of Daily Living scale for use in patients with chronic obstructive pulmonary disease. J Bras Pneumol. 2008 Mar;34(3):143-51. doi: 10.1590/s1806-37132008000300004. English, Portuguese. PMID 18392462
- [Background] Kovelis D, Segretti NO, Probst VS, Lareau SC, Brunetto AF, Pitta F. Validation of the Modified Pulmonary Functional Status and Dyspnea Questionnaire and the Medical Research Council scale for use in Brazilian patients with chronic obstructive pulmonary disease. J Bras Pneumol. 2008 Dec;34(12):1008-18. doi: 10.1590/s1806-37132008001200005. English, Portuguese. PMID 19180335
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Skumlien S, Hagelund T, Bjortuft O, Ryg MS. A field test of functional status as performance of activities of daily living in COPD patients. Respir Med. 2006 Feb;100(2):316-23. doi: 10.1016/j.rmed.2005.04.022. Epub 2005 Jun 6. PMID 15941658
- [Background] Pitta F, Troosters T, Probst VS, Spruit MA, Decramer M, Gosselink R. Quantifying physical activity in daily life with questionnaires and motion sensors in COPD. Eur Respir J. 2006 May;27(5):1040-55. doi: 10.1183/09031936.06.00064105. PMID 16707399
- [Background] Demeyer H, Burtin C, Van Remoortel H, Hornikx M, Langer D, Decramer M, Gosselink R, Janssens W, Troosters T. Standardizing the analysis of physical activity in patients with COPD following a pulmonary rehabilitation program. Chest. 2014 Aug;146(2):318-327. doi: 10.1378/chest.13-1968. PMID 24603844
- [Background] Botega NJ, Bio MR, Zomignani MA, Garcia C Jr, Pereira WA. [Mood disorders among inpatients in ambulatory and validation of the anxiety and depression scale HAD]. Rev Saude Publica. 1995 Oct;29(5):355-63. doi: 10.1590/s0034-89101995000500004. Portuguese. PMID 8731275
- [Background] Silva PN, Jardim JR, Costa e Souza GM, Hyland ME, Nascimento OA. Cultural adaptation and reproducibility of the Breathing Problems Questionnaire for use in patients with COPD in Brazil. J Bras Pneumol. 2012 May-Jun;38(3):339-45. doi: 10.1590/s1806-37132012000300009. English, Portuguese. PMID 22782604
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Jones PW, Quirk FH, Baveystock CM. The St George's Respiratory Questionnaire. Respir Med. 1991 Sep;85 Suppl B:25-31; discussion 33-7. doi: 10.1016/s0954-6111(06)80166-6. PMID 1759018
- [Background] Marques AP, Mendes YC, Taddei U, Pereira CA, Assumpcao A. Brazilian-Portuguese translation and cross cultural adaptation of the activities-specific balance confidence (ABC) scale. Braz J Phys Ther. 2013 Mar-Apr;17(2):170-8. doi: 10.1590/S1413-35552012005000072. PMID 23778771
- [Background] Mesquita R, Wilke S, Smid DE, Janssen DJ, Franssen FM, Probst VS, Wouters EF, Muris JW, Pitta F, Spruit MA. Measurement properties of the Timed Up & Go test in patients with COPD. Chron Respir Dis. 2016 Nov;13(4):344-352. doi: 10.1177/1479972316647178. Epub 2016 Jul 8. PMID 27165963
- [Background] Jacome C, Cruz J, Oliveira A, Marques A. Validity, Reliability, and Ability to Identify Fall Status of the Berg Balance Scale, BESTest, Mini-BESTest, and Brief-BESTest in Patients With COPD. Phys Ther. 2016 Nov;96(11):1807-1815. doi: 10.2522/ptj.20150391. Epub 2016 Apr 14. PMID 27081201
- [Background] Camargos FF, Dias RC, Dias JM, Freire MT. Cross-cultural adaptation and evaluation of the psychometric properties of the Falls Efficacy Scale-International Among Elderly Brazilians (FES-I-BRAZIL). Rev Bras Fisioter. 2010 May-Jun;14(3):237-43. English, Portuguese. PMID 20730369
- [Background] Vincent E, Sewell L, Wagg K, Deacon S, Williams J, Singh S. Measuring a change in self-efficacy following pulmonary rehabilitation: an evaluation of the PRAISE tool. Chest. 2011 Dec;140(6):1534-1539. doi: 10.1378/chest.10-2649. Epub 2011 Jul 7. PMID 21737490
- [Background] Wigal JK, Creer TL, Kotses H. The COPD Self-Efficacy Scale. Chest. 1991 May;99(5):1193-6. doi: 10.1378/chest.99.5.1193. PMID 2019177
- [Background] VLACHOPOULOS, S. P.; NTOUMANIS, N.; SMITH, A. L. The Basic Psychological Needs in Exercise Scale: Translation and evidence for cross-cultural validity. International Journal of Sport and Exercise Psychology, v. 8, p. 394-412, 2010.
- [Background] SCHWARZER, R.; JERUSALÉM, M. Generalized Self-Efficacy scale. In: WEINMAN, J. e WRIGHT, M. J. Measures in health psychology: A user's portfolio. . Windsor, UK: NFER-NELSON, 1995.
- [Background] MARKLAND, D.; TOBIN, V. A. A modification to the Behavioural Regulation in Exercise Questionnaire to include an assessment of amotivation. Journal of Sport and Exercise Psychology, v. 26, n. 2, p. 191-96, 2004.